CLINICAL TRIAL: NCT06799351
Title: Evaluation of the Gut Microbiome Profiles in Patients with Chemotherapy-induced Peripheral Neuropathy Treated in the Randomized Clinical Trial with Ozone OzoParQT (NCT06706544).
Brief Title: Gut Microbiome Profiles in Patients with Chemotherapy-induced Neuropathy in the RCT OzoParQT (NCT06706544).
Acronym: OzoParQTmicrob
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other); Instituto de Salud Carlos III (Other Government); Council of Gran Canaria (Other); CIBER (Infectious diseases) (Unknown); Instituto Universitario de Enfermedades Tropicales y Salud Pública de Canarias, Universidad de La Laguna (Unknown)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, Bernardino Clavo, MD, PhD, Dr. Negrin University Hospital, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 2024-385-1; PIFIISC24/37 (Other Grant/Funding Number: Fundación Canaria Instituto Investigación Sanitaria de Canarias (FIISC)); PI23/01324 (Other Grant/Funding Number: Instituto de Salud Carlos III); CIGC'23/24 (Other Grant/Funding Number: Cabildo de Gran Canaria)
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN); Paresthesia; Numbness; Tingling
Keywords: Chemotherapy induced peripheral neuropathy; paresthesia; numbness and tingling; side effect of cancer treatment; toxicity of chemotherapy; ozone therapy; quality of life; anxiety; depression; oxidative stress; gut microbiota
MeSH Terms: conditions — Paresthesia; Hypesthesia; Anxiety Disorders; Depression | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: This observational study will analyze data from patients enrolled in the randomized, triple-blind, placebo-controlled OzoParQT clinical trial (NCT06706544).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * the oncologists/hematologists who treat and follow the patient regularly,
  * researchers who carry out biochemical determinations or functional tests,
  * researchers who carry out the gut microbiome analysis,
  * statisticians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ozone Group (Experimental): Drug: Ozone (O3/O2). Treatment: Usual treatment + Ozone therapy by rectal insufflation. O3/O2 concentration progressively increased from 10 to 30 μg/ml; 40 sessions in 16 weeks.
  Interventions: Drug: Ozone therapy
- Oxygen Group (Placebo) (Placebo Comparator): Drug: Oxygen (O2). Treatment: Usual treatment + Oxygen by rectal insufflation. O3/O2 concentration = 0 μg/ml (only O2); 40 sessions in 16 weeks.
  Interventions: Drug: Oxygen (placebo)

INTERVENTIONS:
Drug: Ozone therapy — Usual treatment (by their oncologist or hematologist) + Ozone therapy by rectal insufflation. O3/O2 concentration progressively increased from 10 to 30 μg/ml; 40 sessions in 16 weeks.
  Other Names: Ozone treatment; O3/O2 gas mixture; O3
  Arms: Ozone Group
Drug: Oxygen (placebo) — Usual treatment (by their oncologist or hematologist) + Oxygen by rectal insufflation. O3/O2 concentration = 0 μg/ml (only O2); 40 sessions in 16 weeks.
  Other Names: O2
  Arms: Oxygen Group (Placebo)

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common and debilitating side effect of chemotherapy (CT), often requiring dose reductions or treatment interruptions, which can compromise efficacy of the planned CT (limiting its efficacy). Additionally, CIPN usually decreases patients' quality of life.

Unfortunately, effective treatments for CIPN are limited. Emerging evidence suggests potential benefits of rectal ozone therapy and points to a possible role of the gut microbiome in CIPN development and treatment response.

This observational study, ancillary to the randomized clinical trial (RCT) OzoParQT (NCT06706544), investigates the relationship between gut microbiome composition and CIPN severity in patients receiving rectal ozone therapy.

Primary Objectives:

To evaluate if gut microbiome profiles differ between patients:

1. with and without symptomatic improvement of CIPN.
2. receiving rectal ozone therapy and those receiving placebo.

Secondary Objectives:

To evaluate the relationship between gut microbiome composition and:

1. Health-related quality of life,
2. Anxiety and depression,
3. Biochemical markers of oxidative stress and inflammation.

Main Trial Endpoints.

Changes from baseline at the end of ozone therapy (week 16) in:

* Gut microbiome profile
* Patient-reported numbness and tingling
* Neuropathy severity (QLQ-CIPN20 scale)
* Paresthesia toxicity grade (CTCAE v.5.0)

Secondary Trial Endpoints.

Changes from baseline at the end of ozone therapy (week 16) in:

* Patient-reported quality of life (EQ-5D-5L questionnaire)
* Quality of life (QLQ-C30 questionnaire)
* Anxiety and depression levels (HADS questionnaire)
* Biochemical markers of oxidative stress
* Biochemical markers of inflammation

Trial Design:

This observational study will analyze data from patients enrolled in the randomized, triple-blind, placebo-controlled OzoParQT clinical trial (NCT06706544).

Trial Population in the OzoParQT trial (NCT06706544):

Adults (≥18 years) with any tumor type, experiencing CIPN-related paresthesias (numbness and/or tingling), with a toxicity grade ≥ 2 according to the Common Terminology Criteria for Adverse Events (CTCAE v.5.0) for ≥ 3 months.

Intervention in the OzoParQT trial (NCT06706544).

All patients will receive standard care for their CIPN symptoms plus 40 sessions of rectal insufflation of an O3/O2 gas mixture over 16 weeks:

* Ozone group: O3/O2 concentration increasing from 10 to 30 µg/mL
* Control-placebo group: O2 only (0 µg/mL O3)

Study Duration:

Each patient will participate in this study (OzoParQTmicrob) for 16 weeks, concurrent with the ozone therapy intervention. The total planned project duration is 60 months.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common and debilitating side effect of chemotherapy (CT), often requiring dose reductions or treatment interruptions, which can compromise efficacy of the planned CT (limiting its efficacy). Additionally, CIPN usually decreases patients' quality of life.

Unfortunately, effective treatments for CIPN are limited. Emerging evidence suggests potential benefits of rectal ozone therapy and points to a possible role of the gut microbiome in CIPN development and treatment response.

This observational study, ancillary to the randomized clinical trial (RCT) OzoParQT (NCT06706544), investigates the relationship between gut microbiome composition and CIPN severity in patients receiving rectal ozone therapy.

Primary Objectives:

To evaluate if gut microbiome profiles differ between patients:

1. with and without symptomatic improvement of CIPN.
2. receiving rectal ozone therapy and those receiving placebo.

Secondary Objectives:

To evaluate the relationship between gut microbiome composition and:

1. Health-related quality of life,
2. Anxiety and depression,
3. Biochemical markers of oxidative stress and inflammation.

Main Trial Endpoints.

Changes from baseline at the end of ozone therapy (week 16) in:

* Gut microbiome profile
* Patient-reported numbness and tingling
* Neuropathy severity (QLQ-CIPN20 scale)
* Paresthesia toxicity grade (CTCAE v.5.0)

Secondary Trial Endpoints.

Changes from baseline at the end of ozone therapy (week 16) in:

* Patient-reported quality of life (EQ-5D-5L questionnaire)
* Quality of life (QLQ-C30 questionnaire)
* Anxiety and depression levels (HADS questionnaire)
* Biochemical markers of oxidative stress
* Biochemical markers of inflammation

Trial Design:

This observational study will analyze data from patients enrolled in the randomized, triple-blind, placebo-controlled OzoParQT clinical trial (NCT06706544).

Trial Population in the OzoParQT trial (NCT06706544):

Adults (≥18 years) with any tumor type, experiencing CIPN-related paresthesias (numbness and/or tingling), with a toxicity grade ≥ 2 according to the Common Terminology Criteria for Adverse Events (CTCAE v.5.0) for ≥ 3 months.

Intervention in the OzoParQT trial (NCT06706544).

All patients will receive standard care for their CIPN symptoms plus 40 sessions of rectal insufflation of an O3/O2 gas mixture over 16 weeks:

* Ozone group: O3/O2 concentration increasing from 10 to 30 µg/mL
* Control-placebo group: O2 only (0 µg/mL O3)

Study Duration:

Each patient will participate in this study (OzoParQTmicrob) for 16 weeks, concurrent with the ozone therapy intervention. The total planned project duration is 60 months.

ELIGIBILITY:
Inclusion Criteria:

* 0. Patients who agree to participate in the randomized clinical trial OzoParQT, and who also agree to participate in this study of gut microbiota by providing stool samples.
* 1. Adults > = 18 years old.
* 2. Previous treatment with any chemotherapy because of any tumor.
* 3. Clinical diagnosis of paresthesia (numbness, tingling) secondary to CIPN, with toxicity Grade > = 2 (according to the Common Toxicity Criteria for Adverse Events (CTCAE) from the National Cancer Institute of EEUU, v.5.0) for > = 3 months.
* 4. Without neurotoxic chemotherapy > = 3 months.
* 5. Cancer disease is stable or in remission.
* 6. Life expectancy > = 6 months.
* 7. Before enrollment, women of childbearing potential should obtain a negative result in the serum or urine pregnancy test at the screening visit and accept the use of appropriate contraceptive methods at least from 14 days before the first ozone therapy session up to 14 days after the last one.
* 8. To sign and date the specific informed consent of both studies (OzoParQT and OzoParQTmicrob)

Exclusion Criteria:

* 1. Age < 18 years.
* 2. A woman who is lactating, pregnant, suspected of being pregnant, or a woman of childbearing potential who does not use adequate contraceptive methods.
* 3. Suspected symptoms are due to diabetic or compressive neuropathy.
* 4. Severe psychiatric disorders.
* 5. Inability to complete the quality of life questionnaires.
* 6. Elevation above 5 times the maximum limit of normal creatinine.
* 7. Patient who is hemodynamic or clinically unstable or who requires urgent or short-term interventional measures.
* 8. Neoplasia in progression requiring recent initiation of systemic treatment or maintenance with neurotoxic chemotherapy.
* 9. Life expectancy (for any reason) < 6 months.
* 10. Known allergy to ozone, known glucose 6 phosphate dehydrogenase (G6PD) deficiency, or hemochromatosis.
* 11. Contraindications or impossibility for rectal ozone treatment or to attend regularly to the treatment.
* 12. Not meeting each and every one of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in gut microbiome profile, at the end of ozone therapy. | 16 weeks.
  Analysis of gut microbiome profile at the end of ozone therapy regarding the basal profile.
Change from baseline in "numbness and tingling" self-perceived by patients at the end of ozone treatment. | 16 weeks.
  Self-reported evaluation of the percentage of "numbness and/or tingling" regarding the basal level. From 100% (basal level, 0% improvement) to 0% (no numbness and tingling, 100% improvement).
Changes from baseline in the degree of neuropathy according to the QLQ-CIPN20 scale at the end of ozone treatment. | 16 weeks.
  Changes from baseline in the degree of neuropathy according to the QLQ-CIPN20 scale at the end of ozone treatment (from the European Organization for Research & Treatment in Cancer (EORTC)). It is evaluated through 20 items grouped into 3 dimensions: sensory, motor, and autonomic. Range: each item is scored from 1 (nothing) to 4 (a lot). The total score for each dimension is transformed into a score from 0 to 100, with 0 being the best possible state and 100 being the worst.
Changes from baseline in the Grade of toxicity of parestesias (numbness, tingling) according to the CTCAE v.5.0. scale at the end of ozone treatment. | 16 weeks.
  Changes from baseline in the Grade of toxicity of paresthesias (numbness, tingling) according to the CTCAE v.5.0. scale (from the National Cancer Institute of EEUU). Range from: Grade = (asymptomatic or mild symptoms) to Grade 3 (severe symptoms, limiting self-care activities in daily life).

SECONDARY OUTCOMES:
Change from baseline in "Quality of Life" (using the EQ-5D-5L questionnaire) self-perceived by patients at the end of ozone treatment. | 16 weeks.
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (Best: I have no problem) to 5 (worst: I have an extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analog scale (0 = worst health patient can imagine, 100 = best health patient can imagine).
Changes from baseline in the "Quality of Life" according to the QLQ-C30 questionnaire at the end of ozone treatment. | 16 weeks.
  Changes from baseline in the "Quality of Life" according to the QLQ-C30 questionnaire (from the European Organization for Research & Treatment in Cancer (EORTC)). Self-reported evaluation of 30 items that measure several scales and symptoms. Range (after standardization): from 0 (worst for overall health and function, best for symptoms) to 100 (best for overall health and functions, worst for symptoms).
Changes from baseline in levels of anxiety and depression according to the Hospital Anxiety and Depression Scale (HADS), at the end of ozone treatment. | 16 weeks.
  Changes from baseline in levels of anxiety and depression according to the Hospital Anxiety and Depression Scale (HADS). HADS is a self-administered questionnaire that assesses 14 items/symptoms of anxiety (7) and depression (7) experienced by patients. Each item is scored from 0 (better, no alteration) to 3 (worse level of alteration). For each symptom (anxiety or depression), the overall score is from 0 (better, no anxiety or depression) to 21 (worse, very severe anxiety or depression).
Changes from baseline in biochemical parameters of oxidative stress at the end of ozone treatment. | 16 weeks.
  Changes in serum levels of superoxide dismutase, glutathione, glutathione peroxidase and free radicals.
Changes from baseline in biochemical parameters of inflammation at the end of ozone treatment. | 16 weeks.
  Changes in serum levels of pro-inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain; Francisco Rodríguez-Esparragón, BSc, PhD, Study Director — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain; Jacob Lorenzo-Morales, Prof, Principal Investigator — Instituto Universitario de Enfermedades Tropicales y Salud Publica de Canarias - Universidad de La Laguna (IUETSPC-ULL); Francisco Rodríguez-Esparragón, BSc, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain; Bernardino Clavo, MD, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain
Locations (1):
- Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Yes
It will be available (after request):
  * Individual participant data (IPD) that underlie the results reported in further articles, after deidentification
  * Data will be available after publication, ending 36 months following article publication.
  * They will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  * Study protocol
  Proposals should be directed to: bernardinoclavo@gmail.com To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication, ending 36 months following article publication.
Access Criteria: Data will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  - Study protocol
  Proposals should be directed to: bernardinoclavo@gmail.com To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Ramakrishna C, Corleto J, Ruegger PM, Logan GD, Peacock BB, Mendonca S, Yamaki S, Adamson T, Ermel R, McKemy D, Borneman J, Cantin EM. Dominant Role of the Gut Microbiota in Chemotherapy Induced Neuropathic Pain. Sci Rep. 2019 Dec 30;9(1):20324. doi: 10.1038/s41598-019-56832-x. PMID 31889131
- [Background] Lin B, Wang Y, Zhang P, Yuan Y, Zhang Y, Chen G. Gut microbiota regulates neuropathic pain: potential mechanisms and therapeutic strategy. J Headache Pain. 2020 Aug 17;21(1):103. doi: 10.1186/s10194-020-01170-x. PMID 32807072
- [Background] Clavo B, Rodriguez-Abreu D, Galvan-Ruiz S, Federico M, Canovas-Molina A, Ramallo-Farina Y, Antonilli C, Benitez G, Fabelo H, Garcia-Lourve C, Gonzalez-Beltran D, Jorge IJ, Rodriguez-Esparragon F, Callico GM. Long-Term Effects of Ozone Treatment in Patients with Persistent Numbness and Tingling Secondary to Chemotherapy-Induced Peripheral Neuropathy. A Retrospective Study. Integr Cancer Ther. 2025 Jan-Dec;24:15347354241307038. doi: 10.1177/15347354241307038. PMID 39797612
- [Background] Bocci V, Borrelli E, Travagli V, Zanardi I. The ozone paradox: ozone is a strong oxidant as well as a medical drug. Med Res Rev. 2009 Jul;29(4):646-82. doi: 10.1002/med.20150. PMID 19260079
- [Background] Bocci V, Valacchi G. Nrf2 activation as target to implement therapeutic treatments. Front Chem. 2015 Feb 2;3:4. doi: 10.3389/fchem.2015.00004. eCollection 2015. PMID 25699252
- [Background] Bocci VA, Zanardi I, Travagli V. Ozone acting on human blood yields a hormetic dose-response relationship. J Transl Med. 2011 May 17;9:66. doi: 10.1186/1479-5876-9-66. PMID 21575276
- [Background] Clavo B, Canovas-Molina A, Diaz-Garrido JA, Canas S, Ramallo-Farina Y, Laffite H, Federico M, Rodriguez-Abreu D, Galvan S, Garcia-Lourve C, Gonzalez-Beltran D, Carames MA, Hernandez-Fleta JL, Serrano-Aguilar P, Rodriguez-Esparragon F. Effects of ozone therapy on anxiety and depression in patients with refractory symptoms of severe diseases: a pilot study. Front Psychol. 2023 Aug 4;14:1176204. doi: 10.3389/fpsyg.2023.1176204. eCollection 2023. PMID 37599784
- [Background] Clavo B, Canovas-Molina A, Ramallo-Farina Y, Federico M, Rodriguez-Abreu D, Galvan S, Ribeiro I, Marques da Silva SC, Navarro M, Gonzalez-Beltran D, Diaz-Garrido JA, Cazorla-Rivero S, Rodriguez-Esparragon F, Serrano-Aguilar P. Effects of Ozone Treatment on Health-Related Quality of Life and Toxicity Induced by Radiotherapy and Chemotherapy in Symptomatic Cancer Survivors. Int J Environ Res Public Health. 2023 Jan 13;20(2):1479. doi: 10.3390/ijerph20021479. PMID 36674232
- [Background] Clavo B, Martinez-Sanchez G, Rodriguez-Esparragon F, Rodriguez-Abreu D, Galvan S, Aguiar-Bujanda D, Diaz-Garrido JA, Canas S, Torres-Mata LB, Fabelo H, Tellez T, Santana-Rodriguez N, Fernandez-Perez L, Marrero-Callico G. Modulation by Ozone Therapy of Oxidative Stress in Chemotherapy-Induced Peripheral Neuropathy: The Background for a Randomized Clinical Trial. Int J Mol Sci. 2021 Mar 10;22(6):2802. doi: 10.3390/ijms22062802. PMID 33802143
- [Background] Clavo B, Rodriguez-Abreu D, Galvan S, Federico M, Martinez-Sanchez G, Ramallo-Farina Y, Antonelli C, Benitez G, Rey-Baltar D, Jorge IJ, Rodriguez-Esparragon F, Serrano-Aguilar P. Long-term improvement by ozone treatment in chronic pain secondary to chemotherapy-induced peripheral neuropathy: A preliminary report. Front Physiol. 2022 Aug 30;13:935269. doi: 10.3389/fphys.2022.935269. eCollection 2022. PMID 36111149
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Ozone Therapy in Refractory Pelvic Pain Syndromes Secondary to Cancer Treatment: A New Approach Warranting Exploration. J Palliat Med. 2021 Jan;24(1):97-102. doi: 10.1089/jpm.2019.0597. Epub 2020 May 5. PMID 32379556
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Long-Term Results with Adjuvant Ozone Therapy in the Management of Chronic Pelvic Pain Secondary to Cancer Treatment. Pain Med. 2021 Sep 8;22(9):2138-2141. doi: 10.1093/pm/pnaa459. No abstract available. PMID 33738491
- [Background] Clavo B, Rodriguez-Esparragon F, Rodriguez-Abreu D, Martinez-Sanchez G, Llontop P, Aguiar-Bujanda D, Fernandez-Perez L, Santana-Rodriguez N. Modulation of Oxidative Stress by Ozone Therapy in the Prevention and Treatment of Chemotherapy-Induced Toxicity: Review and Prospects. Antioxidants (Basel). 2019 Nov 26;8(12):588. doi: 10.3390/antiox8120588. PMID 31779159
- [Background] Galie M, Covi V, Tabaracci G, Malatesta M. The Role of Nrf2 in the Antioxidant Cellular Response to Medical Ozone Exposure. Int J Mol Sci. 2019 Aug 17;20(16):4009. doi: 10.3390/ijms20164009. PMID 31426459
- [Background] Hidalgo-Tallon J, Menendez-Cepero S, Vilchez JS, Rodriguez-Lopez CM, Calandre EP. Ozone therapy as add-on treatment in fibromyalgia management by rectal insufflation: an open-label pilot study. J Altern Complement Med. 2013 Mar;19(3):238-42. doi: 10.1089/acm.2011.0739. Epub 2012 Oct 9. PMID 23046293
- [Background] Szklener K, Rudzinska A, Juchaniuk P, Kabala Z, Mandziuk S. Ozone in Chemotherapy-Induced Peripheral Neuropathy-Current State of Art, Possibilities, and Perspectives. Int J Mol Sci. 2023 Mar 9;24(6):5279. doi: 10.3390/ijms24065279. PMID 36982352
- [Background] Tricarico G, Travagli V. The Relationship between Ozone and Human Blood in the Course of a Well-Controlled, Mild, and Transitory Oxidative Eustress. Antioxidants (Basel). 2021 Dec 4;10(12):1946. doi: 10.3390/antiox10121946. PMID 34943049
- [Background] Viebahn-Haensler R, Leon Fernandez OS. Ozone in Medicine. The Low-Dose Ozone Concept and Its Basic Biochemical Mechanisms of Action in Chronic Inflammatory Diseases. Int J Mol Sci. 2021 Jul 23;22(15):7890. doi: 10.3390/ijms22157890. PMID 34360655